CLINICAL TRIAL: NCT04812223
Title: Prospective Randomized Comparison of the Results of Early Clamping, Delayed Clamping and Milking of the Umbilical Cord in Term Cesarean Deliveries
Brief Title: Timing of Umbilical Cord Clamping in Term Cesarean Deliveries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Esra Ozbasli, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK 2021-01/44
Record Dates: First submitted 2021-03-17; First posted 2021-03-23 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Cesarean Delivery; Delayed Separation of Umbilical Cord
Keywords: Cesarean delivery; Umbilical cord clamping; Delayed umbilical cord clamping
MeSH Terms: interventions — Umbilical Cord Clamping

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Delayed Clamping (Active Comparator): In this group, the umbilical cord will be clamped 60 seconds after the baby is born.
  Interventions: Procedure: Delayed umbilical cord clamping
- Early Clamping (Active Comparator): In this group, the umbilical cord will be clamped 15 seconds after the baby is born.
  Interventions: Procedure: Early umbilical cord clamping
- Milking Clamping (Active Comparator): In this group in which the umbilical cord will be milked, the cord will be milked 5 times with 2 seconds milking, then letting 2 seconds for spontaneous blood flow.
  Interventions: Procedure: Milking of the umbilical cord

INTERVENTIONS:
Procedure: Delayed umbilical cord clamping — The umbilical cord will be clamped 60 seconds after the baby is born.
  Arms: Delayed Clamping
Procedure: Early umbilical cord clamping — The umbilical cord will be clamped 15 seconds after the baby is born.
  Arms: Early Clamping
Procedure: Milking of the umbilical cord — The cord will be milked 5 times with 2 seconds milking, then letting 2 seconds for spontaneous blood flow.
  Arms: Milking Clamping

SUMMARY:
The aim of this study is to show that delayed umbilical cord clamping or milking of the umbilical cord in pregnant women undergoing elective cesarean delivery might have better effects than early clamping, on neonatal results without causing maternal hemorrhage or negatively affecting the neonatal outcome , and to compare the superiority of these three methods to each other.

DETAILED DESCRIPTION:
Late clamping of the umbilical cord has been shown to have positive effects such as higher neonatal hemoglobin level, higher iron stores in the newborn around three to six months, and better neurological development. In 2017, American College of Obstetricians and Gynecologists (ACOG) recommended a minimum 30-60 seconds delayed clamping of the cord after a minimum of 30-60 seconds, regardless of the delivery method, in both term and preterm newborns. In addition, optimal placental transfusion can be achieved due to strong uterine tonus in vaginal delivery. However, this is not possible due to decreased uterine tonus and time constraint in cesarean delivery. The main concern in delayed clamping and milking of the umbilical cord is the possibility of maternal anemia due to excessive maternal blood loss in the short term, the need for maternal blood transfusion or maternal intensive care support, and the possibility of conditions such as hyperbilirubinemia, symptomatic polycythemia, and long hospital stay that may cause the need for phototherapy in the newborn. Although there are many studies in the literature regarding the neonatal results of the clamping timing of the umbilical cord, there are a limited number of articles regarding the results in patients who underwent term elective cesarean section. The aim of this study is to show that delayed umbilical cord clamping or milking of the umbilical cord in pregnant women undergoing elective cesarean delivery might have better effects than early clamping, on neonatal results without causing maternal hemorrhage or negatively affecting the neonatal outcome , and to compare the superiority of these three methods to each other.

ELIGIBILITY:
Inclusion Criteria:

* > 37 weeks uncomplicated singleton pregnancy
* Elective cesarean delivery
* Cesarean section under regional anesthesia

Exclusion Criteria:

* < 37 weeks pregnancy
* Surgery performed under general anesthesia
* Emergent cesarean
* Multiple pregnancy
* Medically unstable mother or fetus
* Uncontrolled maternal diabetes
* Major congenital malformation of chromosomal abnormality of the fetus
* Intrauterine growth retardation
* Prenatal asphyxia suspicion
* True knot in the umbilical cord
* İn case of meconium aspiration syndrome suspicion

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 204 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-07-25 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Postpartum maternal hemorrhage | On postoperative day 0 and day 2
  Preoperative and postoperative hemoglobin values will be recorded.

SECONDARY OUTCOMES:
Postpartum maternal anemia | İn postpartum 48 hours
  Blood loss during surgery, need for blood transfusion after surgery will be recorded.
Neonatal outcomes | Postpartum day 0
  Weight of the baby
Postpartum complaints | İn postpartum 48 hours
  Postpartum nausea, vomiting, headache, dyspnea will be recorded
Neonatal anemia | On postpartum day 2
  Hematocrit levels of the newborn will be measured
Neonatal jaundice | On postpartum day 2
  Bilirubin levels of the newborn will be measured.
Neonatal intensive care unit admission | In postpartum 5 days
  Neonatal intensive care unit admissions in postpartum 5 days will be recorded.
Maternal outcomes | On postpartum day 2
  Postpartum maternal blood pressure, pulse will be recorded
Newborn phototherapy need | In postpartum 2 weeks
  Need of newborn phototherapy in postpartum 2 weeks will be recorded.
Newborn positive pressure ventilation | Postpartum 5 days
  Need of newborn positive pressure ventilation in postpartum 5 days will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Mete Gungor, MD, Prof., Study Director — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acibadem Maslak Hospital, Istanbul, Sariyer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study protocol, statistical analysis might be shared when the study is completed upon request.

REFERENCES:
- [Background] Committee Opinion No. 684: Delayed Umbilical Cord Clamping After Birth. Obstet Gynecol. 2017 Jan;129(1):1. doi: 10.1097/AOG.0000000000001860. PMID 28002310
- [Background] Mercer JS, Erickson-Owens DA. Rethinking placental transfusion and cord clamping issues. J Perinat Neonatal Nurs. 2012 Jul-Sep;26(3):202-17; quiz 218-9. doi: 10.1097/JPN.0b013e31825d2d9a. PMID 22843002
- [Background] McDonald SJ, Middleton P, Dowswell T, Morris PS. Effect of timing of umbilical cord clamping of term infants on maternal and neonatal outcomes. Cochrane Database Syst Rev. 2013 Jul 11;2013(7):CD004074. doi: 10.1002/14651858.CD004074.pub3. PMID 23843134
- [Background] Songthamwat M, Witsawapaisan P, Tanthawat S, Songthamwat S. Effect of Delayed Cord Clamping at 30 Seconds and 1 Minute on Neonatal Hematocrit in Term Cesarean Delivery: A Randomized Trial. Int J Womens Health. 2020 Jun 23;12:481-486. doi: 10.2147/IJWH.S248709. eCollection 2020. PMID 32607000
- [Background] Purisch SE, Ananth CV, Arditi B, Mauney L, Ajemian B, Heiderich A, Leone T, Gyamfi-Bannerman C. Effect of Delayed vs Immediate Umbilical Cord Clamping on Maternal Blood Loss in Term Cesarean Delivery: A Randomized Clinical Trial. JAMA. 2019 Nov 19;322(19):1869-1876. doi: 10.1001/jama.2019.15995. PMID 31742629
- [Background] Qian Y, Ying X, Wang P, Lu Z, Hua Y. Early versus delayed umbilical cord clamping on maternal and neonatal outcomes. Arch Gynecol Obstet. 2019 Sep;300(3):531-543. doi: 10.1007/s00404-019-05215-8. Epub 2019 Jun 15. PMID 31203386